CLINICAL TRIAL: NCT07207746
Title: Effect of Music on Pain, Embarrassment, and Urodynamic Outcomes During Urodynamic Testing: A Randomized Controlled Trial
Brief Title: Effect of Music on Pain, Embarrassment, and Urodynamic Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, YASEMİN ÖZHANLI, Assist Prof, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024/01.03
Record Dates: First submitted 2025-09-17; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Nursing Care; Pain; Music Intervention
Keywords: music intervention; pain; embarrassment; urodynamic testing
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The study was conducted experimentally with a pre-test and post-test control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinding was used in the study. For this purpose, the participants were not specified in which group they belonged to the research. Therefore, a separate informed consent form was prepared for each group. In order to avoid bias in the analysis of the research data, statistician blinding was also applied.
  While coding the research data, the research groups were coded as A and B, and the statistician was prevented from knowing which letter represented which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Arm (Experimental): Participants in this group listened to slow-tempo (60-80 beats/min) instrumental classical music at a sound level of 40-60 dB throughout the urodynamic procedure (average 30 minutes). Music was delivered via headphones, starting before uroflowmetry and continuing until the end of voiding cystometry. Standard multi-channel urodynamic testing was performed according to the International Continence Society (ICS) Good Urodynamic Practice Guidelines. An 8 Fr cystometry catheter was inserted into the bladder to measure intravesical pressure, and a 4.5 Fr rectal catheter was used to measure intra-abdominal pressure. Urodynamic parameters including bladder capacity, leakage point pressure, detrusor contraction, maximum flow rate (Qmax), detrusor pressure at maximum flow (PdetQmax), and post-void residual volume were recorded. Pain and embarrassment were assessed at three time points: uroflowmetry, sitting on the table, and catheter insertion.
  Interventions: Behavioral: Behavioral: Music Listening
- Control Arm (No Intervention): Participants in this group received standard care during the urodynamic procedure. No music intervention was applied. All procedures were performed under identical conditions following ICS Good Urodynamic Practice Guidelines, with the same catheter sizes and positioning protocol. Pain and embarrassment levels were assessed at the same three time points as in the music group. Urodynamic outcomes were recorded in parallel.

INTERVENTIONS:
Behavioral: Behavioral: Music Listening — Participants listened to slow-tempo instrumental classical music (40-60 dB) via headphones during the entire urodynamic procedure.
  Arms: Music Arm

SUMMARY:
Urodynamic testing (UDT) is a diagnostic procedure frequently used to evaluate lower urinary tract dysfunction, including urinary incontinence and voiding difficulties. Despite its diagnostic value, UDT is invasive and often causes discomfort, pain, and embarrassment due to catheter placement and repeated measurements. These negative experiences may reduce patient compliance, affect diagnostic accuracy, and increase reluctance to repeat the procedure.

Music has been shown to promote relaxation and reduce pain and anxiety in various clinical settings, but its effect during urodynamic testing has not been adequately studied. This randomized controlled trial was designed to determine whether listening to music during invasive UDT can reduce pain and embarrassment while influencing urodynamic parameters.

DETAILED DESCRIPTION:
Urodynamic testing (UDT) is an outpatient diagnostic method used to assess bladder function in patients with lower urinary tract disorders such as urinary incontinence or voiding dysfunction. The procedure involves catheter insertion into the urethra, rectum, or vagina to measure intravesical, detrusor, and urethral pressure, and may include electromyographic evaluation of the external urethral sphincter. UDT typically consists of uroflowmetry, cystometry, and pressure-flow studies, during which urine flow rate and the relationship between intravesical pressure and urine flow are evaluated.

Although essential for diagnosis and treatment planning, UDT is often experienced as stressful and uncomfortable by patients. Pain, embarrassment, and emotional distress are frequently reported due to the invasive nature of catheter placement. These negative experiences may impair patient cooperation, affect the accuracy of urodynamic measurements, and reduce willingness to undergo repeated testing when required for monitoring. Nurses play a key role in preparing and supporting patients during UDT through education, positioning, catheter placement, privacy protection, and emotional support. However, evidence-based complementary strategies to improve patient comfort during UDT remain limited.

Music is a widely recommended nonpharmacological intervention that promotes relaxation, reduces anxiety and pain, and enhances patient satisfaction during invasive procedures. It is safe, cost-effective, and easy to implement. Previous studies have demonstrated that music can improve patient comfort in urological and gastrointestinal procedures, but no randomized controlled trials have specifically investigated its effect during UDT. Considering that patient anxiety and discomfort may influence urination and detrusor function during pressure-flow studies, interventions that improve comfort may also enhance test reliability.

This randomized controlled trial was therefore designed to evaluate the effect of listening to music during invasive urodynamic testing on patient-reported pain, embarrassment, and urodynamic outcomes. The results are expected to contribute to the evidence base for simple, safe, and cost-effective nursing interventions that improve patient comfort and cooperation during UDT.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years who are able to read and write
* Patients scheduled for urodynamic testing
* Patients with no visual, auditory, or cognitive impairments
* Patients without chronic pain

Exclusion Criteria:

* Patients who received sedation during the procedure.
* Pregnant women.
* Patients with a permanent urinary catheter.
* Patients with recurrent or active urinary tract infections.
* Patients requiring urodynamics due to urinary retention.
* Patients with a history of previous urodynamic testing

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Pain Level at Baseline (VAS-P) | T1: 0 minute (before procedure) (Score on a 0-10 scale)
  Pain assessed with a 100 mm VAS (0 = no pain, 10 = worst pain).
Pain Level During Procedure (VAS-P) | T2: 15 minutes (during procedure) (Score on a 0-10 scale)
  Pain assessed with a 100 mm VAS.
Pain Level at End of Procedure (VAS-P) | T3: 30 minutes (end of procedure) (Score on a 0-10 scale)
  Pain assessed with a 100 mm VAS.
Embarrassment Level at Baseline (VAS-E) | T1: 0 minute (before procedure) (Score on a 0-10 scale)
  Embarrassment assessed with a 100 mm VAS (0 = no embarrassment, 10 = maximum embarrassment).
Embarrassment Level During Procedure (VAS-E) | T2: 15 minutes (during procedure) (Score on a 0-10 scale)
  Embarrassment assessed with a 100 mm VAS.
Embarrassment Level at End of Procedure (VAS-E) | T3: 30 minutes (end of procedure) (Score on a 0-10 scale)
  Embarrassment assessed with a 100 mm VAS.

SECONDARY OUTCOMES:
Maximum Flow Rate (Qmax) | Day 1, single measurement during voiding phase (mL/s)
  Maximum urine flow rate recorded during pressure-flow study.
Detrusor Pressure at Maximum Flow (PdetQmax) | Day 1, single measurement during voiding phase (cmH₂O)
  Detrusor pressure measured at maximum urine flow.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, İzmit, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No